CLINICAL TRIAL: NCT03573427
Title: LV Endocardial CRT for Patients With Intermediate QRS Width
Acronym: EndoCRT
Status: Withdrawn | Type: Observational
Why Stopped: No patients enrolled; Executive Committee Decision;Feasibility of recruitment
Sponsor: Jaimie Manlucu (Other)
Responsible Party: Sponsor-Investigator, Jaimie Manlucu, MD, FRCPC, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Other Study IDs: V27Mar17
Record Dates: First submitted 2018-06-05; First posted 2018-06-29 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure，Congestive; Left Ventricular Dysfunction; Left Bundle-Branch Block
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left; Bundle-Branch Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Trans-atrial septal placement LV lead for CRT

SUMMARY:
This pilot study is designed as a multi-centre cohort study determining the degree of LV reverse remodeling in patients with intermediate QRS widths (120-149ms) who undergo CRT implant with transseptal LV leads, and comparing to the average expected reverse remodeling rate in patients with standard transvenous coronary sinus leads and QRS widths ≥150ms.

DETAILED DESCRIPTION:
This is a multi-centre prospective cohort trial to establish the feasibility of endocardial CRT implants.This trial will assess feasibility of a larger scale randomized controlled study.

Patients consented to the study will receive a CRT device with or without ICD, placed in the same time frame, and will have RA and RV leads implanted as the standard of care. The device will be implanted in a facility that has the capacity to perform trans-atrial septal puncture with ultrasound guidance (TEE or ICE) at the time of implantation. The LV lead will be placed using a trans-atrial septal approach, using specially designed puncture tools and LVendo delivery tool kits specifically designed for this study. Special care will be taken to avoid the LV apex and transmural scar identified by pre-implant imaging. Electrical testing, and programming of the device will be standardized.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NYHA Class II-IV ambulatory HF symptoms
* Optimal HF Medical Therapy of at least 3 months (2009 ACCF/AHA, ESC 2012)
* LVEF less than or equal to 35%
* Sinus rhythm (can have paroxysmal atrial fibrillation)
* QRS morphology is non-RBBB
* QRS duration 120-149 ms
* Patients with pacemaker or ICD that meet the above criteria may be upgraded to CRT-D or CRT-P
* Patients are able to receive oral anticoagulation

Exclusion Criteria:

* Patients with atrial septal defect closure
* Planned atrial fibrillation ablation within 12 months
* Patients with mitral prosthetic valve that precludes the placement of an LV lead trans-septally
* Patients with RBBB
* Patients with intra-cardiac thrombi
* Patients with permanent atrial fibrillation
* Patients with contraindications to oral anti-coagulation
* In-hospital patients with acute cardiac or non-cardiac illness that requires intensive care
* Acute coronary syndrome (including MI) < 4 weeks
* Coronary revascularization (CABG or PCI) < 3 months
* Uncorrected or uncorrectable primary valvular disease
* Restrictive, hypertrophic or reversible form of cardiomyopathy
* Severe primary pulmonary disease such as cor pulmonale
* Patients with a life expectancy of less than one year from non-cardiac cause.
* Patients included in other clinical trials that will affect the objectives of this study
* Those unable or unwilling to provide informed consent
* Those with a history of noncompliance to medical therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with left bundle branch block (LBBB) and a QRS width of 120-149 ms; ambulatory NYHA class II-IV heart failure symptoms; and a LV ejection fraction ≤ 35%
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-04-28 (Estimated); Primary Completion 2019-04-28 (Estimated); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
LV end-systolic volume | Change from Baseline measure to 6 months
  Echocardiogram
LVEF improvement | Change from Baseline measure to 6 months
  Echocardiogram

SECONDARY OUTCOMES:
Thromboembolic Events | Through study completion, an average of 1 year
  Adverse Event
Specific system placement procedure related adverse events | Through study completion, an average of 1 year
  Device Implant
Lead(s) dislodgement requiring repositioning or cessation of CRT | Through study completion, an average of 1 year
  Chest xray, device interrogation
Cardiac tamponade requiring intervention | Through study completion, an average of 1 year
  Device Implant
Ventricular Arrhythmias | 6 months, 12 months
  Device interrogation
Mitral Regurgitation | Baseline, 6 months
  Echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Jaimie Manlucu, MD FRCPC, Principal Investigator — Schulich School of Medicine, Western University, London Health Sciences Centre
Locations (8):
- Canada (8):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Science, Halifax, Nova Scotia
  - London Health Science Centre, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Sherbrooke CHUS, Sherbrooke, Quebec